CLINICAL TRIAL: NCT02217475
Title: CENTAUR: Efficacy and Safety Study of Cenicriviroc for the Treatment of Nonalcoholic Steatohepatitis (NASH) in Adult Subjects With Liver Fibrosis
Brief Title: Efficacy and Safety Study of Cenicriviroc for the Treatment of Nonalcoholic Steatohepatitis (NASH) in Adult Participants With Liver Fibrosis
Acronym: CENTAUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 652-2-203; 2016-004754-15 (EudraCT Number)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-03

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — cenicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cenicriviroc (CVC) 150mg/CVC 150 mg (Experimental): CVC 150 mg tablet in Years 1 and 2.
  Interventions: Drug: Cenicriviroc
- Placebo/CVC 150 mg (Experimental): Placebo-matching CVC tablet in Year 1 then CVC 150 mg tablet in Year 2.
  Interventions: Drug: Cenicriviroc; Drug: Placebo
- Placebo/Placebo (Placebo Comparator): Placebo-matching cenicriviroc (CVC) tablet in Years 1 and 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenicriviroc — CVC 150 mg, administered orally once daily and taken every morning with food.
  Other Names: TBR-652
  Arms: Cenicriviroc (CVC) 150mg/CVC 150 mg; Placebo/CVC 150 mg
Drug: Placebo — Placebo administered orally once daily and taken every morning with food.
  Arms: Placebo/CVC 150 mg; Placebo/Placebo

SUMMARY:
The purpose of this study is to determine whether cenicriviroc is effective and safe in the treatment of nonalcoholic steatohepatitis (NASH) in adult participants with liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants aged between 18-75
* Histological evidence of NASH, based on biopsy, with a Nonalcoholic fatty liver disease Activity Score (NAS) of >= 4 with at least 1 in each component of NAS
* Histological evidence of liver fibrosis defined as NASH Clinical Research Network (CRN) System Stage 1 to 3
* Meeting any of the 3 major criteria (a, b, c):

  1. Documented evidence of type 2 diabetes mellitus
  2. High body mass index (> 25 kg/m^2) with at least one of the following criteria of metabolic syndrome, as defined by the National Cholesterol Education Program:

     * Central obesity: waist circumference ≥ 102 cm or 40 inches (male), ≥ 88 cm or 35 inches (female)
     * Dyslipidemia: Triglycerides ≥ 1.7 mmol/L (150 mg/dL)
     * Dyslipidemia: High-density lipoprotein (HDL)-cholesterol < 40 mg/dL (male), < 50 mg/dL (female)
     * Blood pressure ≥ 130/85 mmHg (or currently being treated for hypertension)
     * Fasting plasma glucose ≥ 6.1 mmol/L (110 mg/dL)
  3. Bridging fibrosis (NASH CRN Stage 3) and/or definite NASH (NAS ≥ 5)
* Agree to have one liver biopsy at Screening, one at Year 1, and one at the end of study treatment (Year 2)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × upper limit of normal (ULN)

Exclusion Criteria:

* Hepatitis B surface Antigen (HBsAg) positive
* Hepatitis C antibody (HCVAb) positive with the following 2 exceptions:

  1. Participants previously treated for viral hepatitis C with at least a 1-year period since documented sustained virologic response at Week 12 (post-treatment) may be eligible if all other eligibility criteria are met
  2. Participants with presence of hepatitis C antibody but negative hepatitis C virus ribonucleic acid RNA without treatment (i.e., spontaneous clearance) may be eligible if all other eligibility criteria are met
* Prior or planned liver transplantation
* Other known causes of chronic liver disease, including alcoholic liver disease
* History of cirrhosis and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Alcohol consumption greater than 21 units/week for males or 14 units/week for females (one unit of alcohol is ½ pint of beer [285 mL], 1 glass of spirits [25 mL] or 1 glass of wine [125 mL])
* Human immunodeficiency virus (HIV)-1 or HIV-2 infection
* Weight reduction through bariatric surgery in the past 5 years or planned during the conduct of the study (including gastric banding)
* Females who are pregnant or breastfeeding
* Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with the dosing and protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lefebvre, MD, Study Director — Allergan
Locations (82):
- United States (36):
  - Dothan, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Littleton, Colorado
  - Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Saint Paul, Minnesota
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Buffalo, New York
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Houston, Texas
  - Live Oak, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
- Australia (8):
  - Garran, Australian Capital Territory
  - Herston, Queensland
  - Adelaide, South Australia
  - Bedford Park, South Australia
  - Clayton, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Belgium (3):
  - Brussels
  - Edegem
  - Leuven
- France (8):
  - Angers
  - Lyon
  - Montpellier
  - Paris
  - Pessac
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - Hamburg, Hamburg
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Leipzig, Saxony
  - Heidelberg, VIC
  - Berlin
  - Lübeck
- Shatin, New Territories, Hong Kong
- Italy (4):
  - Bologna, BO
  - Milan, MI
  - Rozzano, MI
  - Palermo, PA
- Poland (5):
  - Chorzów
  - Lodz
  - Mysłowice
  - Rzeszów
  - Wroclaw
- Spain (3):
  - Alicante
  - Barcelona
  - Madrid
- United Kingdom (4):
  - Portsmouth, Hampshire
  - London
  - Newcastle
  - Nottingham

REFERENCES:
- [Derived] Qian T, Fujiwara N, Koneru B, Ono A, Kubota N, Jajoriya AK, Tung MG, Crouchet E, Song WM, Marquez CA, Panda G, Hoshida A, Raman I, Li QZ, Lewis C, Yopp A, Rich NE, Singal AG, Nakagawa S, Goossens N, Higashi T, Koh AP, Bian CB, Hoshida H, Tabrizian P, Gunasekaran G, Florman S, Schwarz ME, Hiotis SP, Nakahara T, Aikata H, Murakami E, Beppu T, Baba H, Rew Warren, Bhatia S, Kobayashi M, Kumada H, Fobar AJ, Parikh ND, Marrero JA, Rwema SH, Nair V, Patel M, Kim-Schulze S, Corey K, O'Leary JG, Klintmalm GB, Thomas DL, Dibas M, Rodriguez G, Zhang B, Friedman SL, Baumert TF, Fuchs BC, Chayama K, Zhu S, Chung RT, Hoshida Y. Molecular Signature Predictive of Long-Term Liver Fibrosis Progression to Inform Antifibrotic Drug Development. Gastroenterology. 2022 Apr;162(4):1210-1225. doi: 10.1053/j.gastro.2021.12.250. Epub 2021 Dec 22. PMID 34951993
- [Derived] Nielsen MJ, Leeming DJ, Goodman Z, Friedman S, Frederiksen P, Rasmussen DGK, Vig P, Seyedkazemi S, Fischer L, Torstenson R, Karsdal MA, Lefebvre E, Sanyal AJ, Ratziu V. Comparison of ADAPT, FIB-4 and APRI as non-invasive predictors of liver fibrosis and NASH within the CENTAUR screening population. J Hepatol. 2021 Dec;75(6):1292-1300. doi: 10.1016/j.jhep.2021.08.016. Epub 2021 Aug 27. PMID 34454994
- [Derived] Parthasarathy G, Malhi H. Macrophage Heterogeneity in NASH: More Than Just Nomenclature. Hepatology. 2021 Jul;74(1):515-518. doi: 10.1002/hep.31790. Epub 2021 May 22. No abstract available. PMID 33666272
- [Derived] Ratziu V, Sanyal A, Harrison SA, Wong VW, Francque S, Goodman Z, Aithal GP, Kowdley KV, Seyedkazemi S, Fischer L, Loomba R, Abdelmalek MF, Tacke F. Cenicriviroc Treatment for Adults With Nonalcoholic Steatohepatitis and Fibrosis: Final Analysis of the Phase 2b CENTAUR Study. Hepatology. 2020 Sep;72(3):892-905. doi: 10.1002/hep.31108. Epub 2020 Jul 21. PMID 31943293
- [Derived] Lefebvre E, Moyle G, Reshef R, Richman LP, Thompson M, Hong F, Chou HL, Hashiguchi T, Plato C, Poulin D, Richards T, Yoneyama H, Jenkins H, Wolfgang G, Friedman SL. Antifibrotic Effects of the Dual CCR2/CCR5 Antagonist Cenicriviroc in Animal Models of Liver and Kidney Fibrosis. PLoS One. 2016 Jun 27;11(6):e0158156. doi: 10.1371/journal.pone.0158156. eCollection 2016. PMID 27347680
- [Derived] Friedman S, Sanyal A, Goodman Z, Lefebvre E, Gottwald M, Fischer L, Ratziu V. Efficacy and safety study of cenicriviroc for the treatment of non-alcoholic steatohepatitis in adult subjects with liver fibrosis: CENTAUR Phase 2b study design. Contemp Clin Trials. 2016 Mar;47:356-65. doi: 10.1016/j.cct.2016.02.012. Epub 2016 Mar 2. PMID 26944023

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 812 participants were screened, and 289 participants were randomized to treatment period 1. Of the 289 participants randomized, 250 participants completed Treatment Period 1. A total of 242 participants entered Treatment Period 2 and 212 completed.
Groups:
- Placebo/Placebo: Placebo-matching cenicriviroc (CVC) tablet, once daily in the morning with food in Years 1 and 2.
- Placebo/Cenicriviroc (CVC) 150 mg: Placebo-matching CVC tablet, once daily in the morning with food in Year 1 then CVC 150 mg tablet, once daily in the morning with food in Year 2.
- CVC 150mg/CVC 150 mg: CVC 150 mg tablet, once daily in the morning with food in Years 1 and 2.
Period: Treatment Period 1 (Year 1)
Arm/Group | Placebo/Placebo | Placebo/Cenicriviroc (CVC) 150 mg | CVC 150mg/CVC 150 mg
Started | 72 | 72 | 145
Safety Analysis Set (Received at least one dose of study drug.) | 72 | 72 | 144
Completed | 62 | 64 | 124
Not Completed | 10 | 8 | 21
Not completed — Protocol Deviation (with non-compliance) | 0 | 1 | 0
Not completed — Adverse Event | 4 | 5 | 9
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Subject Withdrew Consent | 5 | 2 | 11
Not completed — Other Miscellaneous Reasons | 0 | 0 | 1
Period: Discontinued After Period 1
Arm/Group | Placebo/Placebo | Placebo/Cenicriviroc (CVC) 150 mg | CVC 150mg/CVC 150 mg
Started | 62 | 64 | 124
Completed | 60 | 61 | 121
Not Completed | 2 | 3 | 3
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Participant Withdrew Consent | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1
Period: Treatment Period 2 (Year 2)
Arm/Group | Placebo/Placebo | Placebo/Cenicriviroc (CVC) 150 mg | CVC 150mg/CVC 150 mg
Started | 60 | 61 | 121
Completed | 58 | 59 | 109
Not Completed | 2 | 2 | 12
Not completed — Adverse Event | 0 | 1 | 5
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Subject Withdrew Consent | 2 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Other Miscellaneous Reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants regardless of starting treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVC 150mg/CVC 150 mg | Placebo/Cenicriviroc (CVC) 150 mg | Placebo/Placebo | Total
Number analyzed (Participants) | 145 | 72 | 72 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.22) | 55.3 (10.38) | 52.1 (11.37) | 54.1 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 39 | 40 | 152
  Male | 72 | 33 | 32 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 18 | 7 | 48
  Not Hispanic or Latino | 122 | 51 | 65 | 238
  Not reported | 0 | 2 | 0 | 2
  Unknown | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 9 | 21
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Black or African American | 5 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
  White | 129 | 63 | 58 | 250
  Other | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Hepatic Histological Improvement in NAS by ≥ 2 Points With at Least 1-Point Reduction in Either Lobular Inflammation or Hepatocellular Ballooning and no Concurrent Worsening of Fibrosis at Year 1
Description: Hepatic histological improvement in Nonalcoholic Fatty Liver Disease Activity Score (NAS) at Year 1 was defined as a decrease (improvement) in NAS by ≥ 2 with at least a 1-point reduction in either lobular inflammation or hepatocellular ballooning and with no concurrent worsening of fibrosis stage. The NAS was derived as the unweighted sum of steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocellular ballooning (0 to 2) scores. The NAS ranges from 0-8 with the higher score indicating more aggressive disease. Evaluation of fibrosis stage was based on the nonalcoholic steatohepatitis clinical research network (NASH CRN) fibrosis staging system, which was scaled from 0 to 4 stages where, 0=None to 4=Cirrhosis. Worsening of fibrosis stage was defined as progression of NASH CRN fibrosis stage.
Time Frame: Year 1
Population: Intent-to-treat (ITT) population included all randomized participants regardless of starting treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo-matching cenicriviroc tablet, once daily in the morning with food in Year 1.
- CVC 150 mg: Cenicriviroc 150 mg tablet, once daily in the morning with food in Year 1.
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 145
Participants | 27 | 23
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.5194, Regression, Logistic; Logistic regression model was used for analysis. Randomized treatment group, NAS score at screening and fibrosis stage were the factors; Odds Ratio (OR) = 0.816, 95% CI 2-sided [0.439 to 1.516]

2. Secondary Outcome: Number of Participants With Complete Resolution of Steatohepatitis With no Concurrent Worsening of Fibrosis Stage and Improvement in Fibrosis by at Least 1 Stage (NASH CRN System) and no Worsening of Steatohepatitis at Year 1
Description: Complete resolution of steatohepatitis was defined as histopathologic interpretation of no fatty liver disease, or simple or isolated steatosis with no steatohepatitis. As per NASH CRN system, no worsening of steatohepatitis was defined as no worsening of lobular inflammation or hepatocellular ballooning grade. The evaluation of fibrosis stage associated with NASH was based on the NASH CRN fibrosis staging system which was scaled from 0 to 4 stages where, 0=None to 4=Cirrhosis.
Time Frame: Year 1
Population: ITT population included all randomized participants regardless of starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 145
Participants | 4 | 7
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.0388, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.934, 95% CI 2-sided [1.035 to 3.614]

3. Secondary Outcome: Number of Participants With Complete Resolution of Steatohepatitis With no Concurrent Worsening of Fibrosis Stage and Improvement in Fibrosis by at Least 1 Stage (NASH CRN System) and no Worsening of Steatohepatitis at Year 2
Description: as for outcome 2
Time Frame: Year 2
Population: ITT population Year 2 included all participants who had an evaluable year 1 biopsy and received at least 1 dose of study drug during Year 2.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo-matching cenicriviroc tablet, once daily in the morning with food in Years 1 and 2.
- CVC 150 mg: Cenicriviroc 150 mg tablet or placebo-matching cenicriviroc tablet, once daily in the morning with food in Year 1 then cenicriviroc 150 mg tablet, once daily in the morning with food in Year 2.
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 57 | 178
Participants | 2 | 5
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.5920, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.249, 95% CI 2-sided [0.553 to 2.821]

4. Secondary Outcome: Number of Participants With Complete Resolution of Steatohepatitis With no Concurrent Worsening of Fibrosis Stage at Year 1
Description: as for outcome 2
Time Frame: Year 1
Population: ITT population included all randomized participants regardless of starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 145
Participants | 8 | 11
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.4941, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.396, 95% CI 2-sided [0.537 to 3.628]

5. Secondary Outcome: Number of Participants With Complete Resolution of Steatohepatitis With no Concurrent Worsening of Fibrosis Stage at Year 2
Description: as for outcome 2
Time Frame: Year 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 57 | 178
Participants | 3 | 11
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.8434, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.142, 95% CI 2-sided [0.305 to 4.277]

6. Secondary Outcome: Number of Participants With Improvement in Fibrosis by at Least 1 Stage (NASH CRN System) and no Worsening of Steatohepatitis at Year 1
Description: The evaluation of fibrosis stage associated with NASH was based on the NASH CRN Fibrosis Staging System which was scaled from 0 to 4 stages where, 0=None to 4=Cirrhosis. As per NASH CRN system, no worsening of steatohepatitis was defined as no worsening of lobular inflammation or hepatocellular ballooning grade.
Time Frame: Year 1
Population: ITT population included all randomized participants regardless of starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 145
Participants | 15 | 29
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.0234, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.201, 95% CI 2-sided [1.113 to 4.352]

7. Secondary Outcome: Number of Participants With Improvement in Fibrosis by at Least 1 Stage (NASH CRN System) and no Worsening of Steatohepatitis at Year 2
Description: as for outcome 6
Time Frame: Year 2
Population: ITT analysis set Year 2 included all participants who have an evaluable year 1 biopsy and who received at least one dose of study drug during Year 2 (after the 1 year biopsy).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 57 | 178
Participants | 8 | 27
Statistical Analysis 1: Comparison: Placebo vs CVC 150 mg; Test type: Superiority; p = 0.7474, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.154, 95% CI 2-sided [0.484 to 2.752]

8. Secondary Outcome: Number of Participants With Deaths, Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), TEAEs Leading Study Drug to Discontinuation
Description: A TEAE was defined as any adverse event that started or worsened on or after the start of the study medication and up to 30 days after the discontinuation of the study medication. An SAE was defined as any untoward medical occurrence that, at any dose, results in death, was life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: Years 1 and 2
Population: Safety Analysis Set Year 1 and Year 2 included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- CVC 150 mg/CVC 150 mg: CVC 150 mg tablet, once daily in the morning with food in Years 1 and 2.
- Placebo/CVC 150 mg: Placebo-matching CVC tablet, once daily in the morning with food in Year 1 then CVC 150 mg tablet, once daily in the morning with food in Year 2.
Arm/Group | CVC 150 mg/CVC 150 mg | Placebo/CVC 150 mg | Placebo/Placebo
Number analyzed (Participants) | 144 | 72 | 72
Participants
  Deaths | 0 | 0 | 0
  TEAEs | 137 | 68 | 70
  SAEs | 25 | 8 | 12
  TEAEs Leading Study Drug to Discontinuation | 14 | 8 | 5

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included blood pressure, temperature, heart rate, and respiration rate. Vital signs were reviewed by the Investigator for clinically significant changes.
Time Frame: Years 1 and 2
Population: Safety Analysis Set Year 1 and Year 2 included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CVC 150 mg/CVC 150 mg | Placebo/CVC 150 mg | Placebo/Placebo
Number analyzed (Participants) | 144 | 72 | 72
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Grade 3-4 abnormal clinical laboratory values that occurred in ≥2% participants were reported. Criteria used for various parameters was:Fasting glucose Grade3:>250 - 500 mg/dL and Grade4: >500 mg/dL; Alanine aminotransferase(ALT)Grade3:>5.0 - 20.0 ×Upper Limit of Normal(ULN)and Grade4:>20.0 ×ULN; Aspartate aminotransferase(AST)Grade3: >5.0 - 20.0 ×ULN and Grade4: >20.0 ×ULN; Activated partial thromboplastin(APT)/Partial thromboplastin time(PTT)Grade3: >2.5×ULN; Triglycerides Grade3 >500 - 1000 mg/dL and Grade4: >1000 mg/dL; Gamma-glutamyl transferase(GGT)Grade3: >5.0 - 20.0 ×ULN and Grade4: >20.0 ×ULN; Creatine kinase Grade 3: >5.0 - 10.0 ×ULN and Grade4: >10.0 ×ULN; Uric acid Grade3:(ULN - 10 mg/dL; ULN - 0.59 mmol/L) and Grade4: >10 mg/dL; Amylase Grade3: >2.0 - 5.0 ×ULN and Grade4: >5.0 ×ULN; Lipase Grade3: >2.0 - 5.0 xULN and Grade4: >5.0 xULN; Phosphorus Grade3: <2.0 - 1.0 mg/dL and Grade4: <1.0 mg/dL and Absolute neutrophil Grade3: <1.0 - 0.5 × 109/L and Grade4: <0.5 × 109/L.
Time Frame: Years 1 and 2
Population: Safety Analysis Set Year 1 and Year 2 included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- CVC 150 mg (Year 1): CVC 150 mg tablet, once daily in the morning with food in Year 1.
- Placebo (Year 1): Placebo-matching cenicriviroc tablet once daily in the morning with food in Year 1.
- Placebo Then CVC 150 mg: Placebo-matching cenicriviroc tablet, once daily in the morning with food in Year 1 then Cenicriviroc 150 mg tablet, once daily in the morning with food in Year 2. Includes AEs that occurred in Year 2.
- Placebo Then Placebo: Placebo-matching cenicriviroc tablet, once daily in the morning with food in Years 1 and 2. Includes AEs that occurred in Year 2.
Arm/Group | CVC 150 mg (Year 1) | Placebo (Year 1) | CVC 150 mg | Placebo Then CVC 150 mg | Placebo Then Placebo
Number analyzed (Participants) | 144 | 144 | 121 | 61 | 60
Participants
  Fasting glucose (Grade 3) | 17 | 13 | 10 | 6 | 5
  Fasting glucose (Grade 4) | 0 | 0 | 0 | 0 | 0
  ALT (Grade 3) | 17 | 17 | 4 | 3 | 2
  ALT (Grade 4) | 0 | 0 | 0 | 0 | 0
  AST (Grade 3) | 7 | 10 | 1 | 3 | 1
  AST (Grade 4) | 0 | 0 | 0 | 0 | 0
  APT/PTT (Grade 3) | 4 | 2 | 1 | 1 | 2
  Triglycerides (Grade 3) | 5 | 7 | 6 | 5 | 2
  Triglycerides (Grade 4) | 3 | 3 | 2 | 0 | 1
  GGT (Grade 3) | 8 | 7 | 8 | 2 | 2
  GGT (Grade 4) | 1 | 1 | 1 | 0 | 0
  Creatine kinase (Grade 3) | 6 | 7 | 1 | 2 | 4
  Creatine kinase (Grade 4) | 2 | 2 | 3 | 1 | 0
  Uric acid (Grade 3) | 9 | 8 | 4 | 3 | 2
  Uric acid (Grade 4) | 11 | 6 | 5 | 1 | 6
  Amylase (Grade 3) | 6 | 1 | 4 | 0 | 1
  Amylase (Grade 4) | 3 | 0 | 2 | 0 | 0
  Lipase (Grade 3) | 4 | 2 | 3 | 0 | 1
  Lipase (Grade 4) | 5 | 0 | 3 | 0 | 1
  Phosphorus (Grade 3) | 5 | 2 | 2 | 1 | 1
  Phosphorus (Grade 4) | 0 | 0 | 0 | 0 | 0
  Absolute neutrophil (Grade 3) | 2 | 3 | 3 | 0 | 1
  Absolute neutrophil (Grade 4) | 2 | 1 | 1 | 1 | 1

11. Secondary Outcome: Number of Participants With Clinically Abnormal in Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was performed. ECG results were reviewed by the Investigator for clinically notable abnormalities.
Time Frame: Years 1 and 2
Population: Safety Analysis Set Year 1 and Year 2 included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CVC 150 mg/CVC 150 mg | Placebo/CVC 150 mg | Placebo/Placebo
Number analyzed (Participants) | 144 | 72 | 72
Participants | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Hepatic Histological Improvement in NAS at Year 2
Description: Hepatic histological improvement in NAS at Year 2 was defined as a decrease (improvement) in NAS by ≥ 2 with at least a 1-point reduction in either lobular inflammation or hepatocellular ballooning and with no concurrent worsening of fibrosis stage. The NAS was derived as the unweighted sum of steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocellular ballooning (0 to 2) scores. The NAS ranges from 0-8 with the higher score indicating more aggressive disease.
Time Frame: Year 2
Population: Full Analysis Set (FAS) in Year 2 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
Participants | 7 | 24

13. Secondary Outcome: Change From Baseline in the 3 Categorical Features of NAS (Steatosis, Lobular Inflammation, Hepatocellular Ballooning) at Year 1
Description: NAS was calculated using the following 3 categorical features: steatosis which was scaled from 0-3 (steatosis score is defined as 0= <5%, 1= 5 - 33%, 2= >33 - 66%, and 3= >66%), lobular inflammation which was scaled from 0-3 (lobular inflammation score defined as 0= no foci, 1= < 2 foci/200x, 2= 2-4 foci/200x, and 3= > 4 foci/200x), and hepatocellular ballooning which was scaled from 0-2 (hepatocellular ballooning score is defined as 0=none, 1=few balloon cells, 2=many cells/prominent ballooning). A negative change from Baseline indicates improvement.
Time Frame: Year 1
Population: FAS in Year 1 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 126 | 126
score on a scale
  Baseline (Steatosis) | 1.4 (0.55) | 1.3 (0.57)
  Change from Baseline (Steatosis) | -0.1 (0.66) | -0.2 (0.56)
  Baseline (Lobular Inflammation) | 2.5 (0.56) | 2.4 (0.58)
  Change from Baseline (Lobular Inflammation) | -0.1 (0.79) | -0.1 (0.88)
  Baseline (Hepatocellular Ballooning) | 1.5 (0.50) | 1.5 (0.50)
  Change from Baseline (Hepatocellular Ballooning) | -0.2 (0.75) | -0.1 (0.75)

14. Secondary Outcome: Change From Baseline in the 3 Categorical Features of NAS (Steatosis, Lobular Inflammation, Hepatocellular Ballooning) at Year 2
Description: as for outcome 13
Time Frame: Year 2
Population: FAS in Year 2 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 54 | 159
score on a scale
  Baseline (Steatosis) | 1.5 (0.54) | 1.3 (0.52)
  Change from Baseline (Steatosis) | -0.4 (0.56) | -0.2 (0.50)
  Baseline (Lobular Inflammation) | 2.4 (0.63) | 2.4 (0.54)
  Change from Baseline (Lobular Inflammation) | 0.1 (0.72) | 0.0 (0.84)
  Baseline (Hepatocellular Ballooning) | 1.5 (0.50) | 1.5 (0.50)
  Change from Baseline (Hepatocellular Ballooning) | -0.1 (0.68) | 0.0 (0.83)

15. Secondary Outcome: Number of Participants With Hepatic Histological Improvement With a Minimum 2-Point Improvement in NAS With at Least a 1-Point Improvement in More Than 1 Categorical Features of NAS and no Concurrent Worsening of Fibrosis Stage at Year 1
Description: Hepatic histological improvement in NAS was defined as a decrease (improvement) in NAS by ≥ 2 with at least a 1-point reduction in either steatosis, lobular inflammation or hepatocellular ballooning and with no concurrent worsening of fibrosis stage. The NAS was derived as the unweighted sum of steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocellular ballooning (0 to 2) scores. The NAS ranges from 0-8 with the higher score indicating more aggressive disease. Worsening was defined as progression of NASH CRN fibrosis stage.
Time Frame: Year 1
Population: FAS in Year 1 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
Participants | 24 | 22

16. Secondary Outcome: Number of Participants With Hepatic Histological Improvement With a Minimum 2-Point Improvement in NAS With at Least a 1-point Improvement in More Than 1 Categorical Features of NAS and no Concurrent Worsening of Fibrosis Stage at Year 2
Description: as for outcome 15
Time Frame: Year 2
Population: FAS in Year 2 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
Participants | 6 | 20

17. Secondary Outcome: Number of Participants With Resolution of NASH Using a Modified Definition Based on Categorical Features of NAS and no Concurrent Worsening of Fibrosis Stage at Year 1
Description: Resolution of NASH was defined as having no hepatocellular ballooning (grade 0) and minimal to no lobular inflammation (grade 1 or 0) with no concurrent worsening of fibrosis stage (worsening defined as progression of NASH CRN fibrosis stage).
Time Frame: Year 1
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
Participants | 7 | 6

18. Secondary Outcome: Number of Participants With Resolution of NASH Using a Modified Definition Based on Categorical Features of NAS and no Concurrent Worsening of Fibrosis Stage at Year 2
Description: as for outcome 17
Time Frame: Year 2
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
Participants | 1 | 9

19. Secondary Outcome: Change From Baseline in Morphometric Quantitative Collagen on Liver Biopsy at Year 1
Description: The morphometric quantitative collagen on liver biopsy was determined as percent collagen area (PCA) using Sirius red stain on liver biopsy at Year 1. A negative change from Baseline indicates improvement.
Time Frame: Year 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent collagen area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 123 | 121
percent collagen area
  Baseline | 2.49 (2.004) | 2.37 (1.827)
  Change from Baseline to Year 1 | -0.14 (2.389) | 0.02 (2.357)

20. Secondary Outcome: Change From Baseline in Morphometric Quantitative Collagen on Liver Biopsy at Year 2
Description: The morphometric quantitative collagen on liver biopsy was determined as percent collagen area (PCA) using Sirius red stain on liver biopsy at Year 2. A negative change from Baseline indicates improvement.
Time Frame: Year 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent collagen area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 51 | 150
percent collagen area
  Baseline | 2.57 (2.156) | 2.48 (1.892)
  Change from Baseline to Year 2 | -0.17 (2.576) | -0.09 (2.160)

21. Secondary Outcome: Change From Baseline in Hepatic Tissue Fibrogenic Protein Alpha-Smooth Muscle Actin (α-SMA) at Year 1
Description: The hepatic tissue fibrogenic protein α-SMA level was determined as percent α-SMA + area using α-SMA stain on liver biopsy at Year 1. A positive change from Baseline indicates worsening.
Time Frame: Baseline (Day 1) to Year 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of α-SMA positive cells/area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 122 | 122
percentage of α-SMA positive cells/area
  Baseline | 2.41 (2.264) | 2.49 (2.885)
  Change from Baseline to Year 1 | 0.77 (3.529) | 0.79 (3.861)

22. Secondary Outcome: Change From Baseline in Hepatic Tissue Fibrogenic Protein Alpha-Smooth Muscle Actin (α-SMA) at Year 2
Description: The hepatic tissue fibrogenic protein α-SMA level was determined as percent α-SMA + area using α-SMA stain on liver biopsy at Year 2. A positive change from Baseline indicates worsening.
Time Frame: Baseline (Day 1) to Year 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage of α-SMA positive cells/area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 52 | 152
percentage of α-SMA positive cells/area
  Baseline | 2.47 (2.679) | 2.44 (2.505)
  Change from Baseline to Year 2 | 2.10 (4.533) | 1.38 (3.793)

23. Secondary Outcome: Change From Baseline in Morphometric Quantitative Fat Content on Liver Biopsy at Year 1
Description: The morphometric quantitative fat content was done to find out the amount of fat accumulated in the liver. A liver biopsy was performed to determine percent fat area, at Year 1. A negative change from Baseline indicates improvement.
Time Frame: Year 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent fat area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 123 | 121
percent fat area
  Baseline | 22.42 (10.016) | 21.58 (8.740)
  Change from Baseline to Year 1 | -3.39 (9.120) | -2.79 (8.127)

24. Secondary Outcome: Change From Baseline in Morphometric Quantitative Fat Content on Liver Biopsy at Year 2
Description: The morphometric quantitative fat content was done to find out the amount of fat accumulated in the liver. A liver biopsy was performed to determine percent fat area, at Year 2. A negative change from Baseline indicates improvement.
Time Frame: Year 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent fat area
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 50 | 150
percent fat area
  Baseline | 23.30 (10.300) | 21.62 (9.575)
  Change from Baseline to Year 2 | -5.06 (9.739) | -2.96 (9.230)

25. Secondary Outcome: Change From Baseline in Histologic Fibrosis Stage (NASH CRN System and Ishak Scale Score) at Year 1
Description: The participant's histologic fibrosis stage was determined using the NASH CRN system and Ishak scale score assessment at Year 1. The evaluation of fibrosis stage associated with NASH was based on the NASH CRN Fibrosis Staging System which was scaled from 0 to 4 where, 0=None to 4=Cirrhosis. The histologic fibrosis stage based on the Ishak assessment was divided into 1 to 6 stages. Fibrosis was staged with the Ishak scale (ranging from 0=No fibrosis to 6=Cirrhosis). A positive change from Baseline indicates worsening.
Time Frame: Baseline (Day 1) to Year 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 126 | 126
score on a scale
  Baseline (NASH CRN Fibrosis Stage) | 2.1 (0.86) | 2.0 (0.85)
  Change from Baseline (NASH CRN Fibrosis Stage) | 0.2 (0.92) | 0.0 (1.00)
  Baseline (Ishak Fibrosis Stage) | 2.2 (1.00) | 2.2 (1.05)
  Change from Baseline (Ishak Fibrosis Stage) | 0.2 (1.10) | 0.0 (1.20)

26. Secondary Outcome: Change From Baseline in Histologic Fibrosis Stage (NASH CRN System and Ishak Scale Score) at Year 2
Description: The participant's histologic fibrosis stage was determined using the NASH CRN system and Ishak scale score assessment at Year 1. The evaluation of fibrosis stage associated with NASH was based on the NASH CRN Fibrosis Staging System which was scaled from 0 to 4 where, 0=None to 4=Cirrhosis. The histologic fibrosis stage based on the Ishak assessment was divided into 1 to 6 stages. Fibrosis was staged with the Ishak scale (ranging from 0=No fibrosis to 6=Cirrhosis). A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Year 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 54 | 159
score on a scale
  Baseline (NASH CRN Fibrosis Stage) | 2.0 (0.88) | 2.1 (0.85)
  Change from Baseline (NASH CRN Fibrosis Stage) | 0.0 (0.89) | 0.0 (1.08)
  Baseline (Ishak Fibrosis Stage) | 2.1 (1.00) | 2.2 (1.04)
  Change from Baseline (Ishak Fibrosis Stage) | 0.1 (1.21) | 0.0 (1.26)

27. Secondary Outcome: Change From Baseline in Portal Inflammation Grade on Liver Biopsy at Year 1
Description: Portal inflammation on liver biopsy was graded from 0 to 4 where 0= None, 1= Mild, 2= Moderate, and 3= Marked. A positive change from Baseline indicates worsening.
Time Frame: Baseline (Day 1) to Year 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 126 | 124
score on a scale
  Baseline | 1.6 (0.63) | 1.5 (0.64)
  Change from Baseline to Year 1 | 0.0 (0.76) | 0.2 (0.74)

28. Secondary Outcome: Change From Baseline in Portal Inflammation Grade on Liver Biopsy at Year 2
Description: as for outcome 27
Time Frame: Baseline (Day 1) to Year 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 54 | 159
score on a scale
  Baseline | 1.5 (0.64) | 1.6 (0.67)
  Change from Baseline to Year 1 | 0.1 (0.75) | 0.2 (0.72)

29. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Aspartate Aminotransferase to Platelet Count Ratio Index (APRI) at Months 3, 6 and 12
Description: APRI is the ratio of aspartate aminotransferase (AST) to platelet count. It is calculated using formula, APRI = (AST level [/ULN] / platelet counts [10^9/L]) * 100. An APRI index of <=0.50 indicated the absence of significant fibrosis and an index of > 1.50 indicated the presence of significant fibrosis. A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline (Month 0) to Months 3, 6 and 12
Population: FAS in Year 1 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations. Number analyzed is the number of participants with data available for analysis at both Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
ratio
  Baseline (Month 3): number analyzed (Participants) | 127 | 133
  Baseline (Month 3) | 0.649 (0.3661) | 0.596 (0.4089)
  Change from Baseline to Month 3: number analyzed (Participants) | 127 | 133
  Change from Baseline to Month 3 | -0.005 (0.3012) | 0.065 (0.3152)
  Baseline (Month 6): number analyzed (Participants) | 128 | 127
  Baseline (Month 6) | 0.663 (0.3811) | 0.578 (0.3794)
  Change from Baseline to Month 6: number analyzed (Participants) | 128 | 127
  Change from Baseline to Month 6 | 0.009 (0.3968) | 0.102 (0.4536)
  Baseline (Month 12): number analyzed (Participants) | 117 | 117
  Baseline (Month 12) | 0.662 (0.3915) | 0.580 (0.3939)
  Change from Baseline to Month 12: number analyzed (Participants) | 117 | 117
  Change from Baseline to Month 12 | 0.066 (0.5572) | 0.093 (0.3852)

30. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Aspartate Aminotransferase to Platelet Count Ratio Index (APRI) at Months 15, 18 and 24
Description: as for outcome 29
Time Frame: Baseline (Month 0) to Months 15, 18 and 24
Population: FAS in Year 2 included all participants who were randomized and received at least 1 dose of study drug, had a measurable Screening biopsy, and had no major eligibility violations. Number analyzed is the number of participants with data available for analysis at both Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
ratio
  Baseline (Month 15): number analyzed (Participants) | 59 | 167
  Baseline (Month 15) | 0.619 (0.3157) | 0.584 (0.3572)
  Change from Baseline to Month 15: number analyzed (Participants) | 59 | 167
  Change from Baseline to Month 15 | 0.002 (0.3422) | 0.118 (0.4095)
  Baseline (Month 18): number analyzed (Participants) | 53 | 167
  Baseline (Month 18) | 0.620 (0.3305) | 0.586 (0.3612)
  Change from Baseline to Month 18: number analyzed (Participants) | 53 | 167
  Change from Baseline to Month 18 | 0.038 (0.4033) | 0.133 (0.4269)
  Baseline (Month 24): number analyzed (Participants) | 56 | 158
  Baseline (Month 24) | 0.633 (0.3156) | 0.584 (0.3617)
  Change from Baseline to Month 24: number analyzed (Participants) | 56 | 158
  Change from Baseline to Month 24 | -0.020 (0.4721) | 0.086 (0.4153)

31. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Fibrosis-4 (FIB-4) at Months 3, 6 and 12
Description: Fibrosis-4 is the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, alanine aminotransferase (ALT), AST and age that is calculated using formula: FIB-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of < 1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis. A positive change from Baseline indicates increased fibrosis.
Time Frame: Baseline (Month 0) to Months 3, 6 and 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
ratio
  Baseline (Month 3): number analyzed (Participants) | 127 | 133
  Baseline (Month 3) | 1.444 (0.6753) | 1.417 (0.6893)
  Change from Baseline to Month 3: number analyzed (Participants) | 127 | 133
  Change from Baseline to Month 3 | 0.021 (0.4236) | 0.071 (0.4209)
  Baseline (Month 6): number analyzed (Participants) | 128 | 127
  Baseline (Month 6) | 1.500 (0.7268) | 1.388 (0.6771)
  Change from Baseline to Month 6: number analyzed (Participants) | 128 | 127
  Change from Baseline to Month 6 | 0.015 (0.4591) | 0.099 (0.5246)
  Baseline (Month 12): number analyzed (Participants) | 117 | 117
  Baseline (Month 12) | 1.503 (0.7442) | 1.398 (0.6834)
  Change from Baseline to Month 12: number analyzed (Participants) | 117 | 117
  Change from Baseline to Month 12 | 0.106 (0.6876) | 0.117 (0.5069)

32. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Fibrosis-4 (FIB-4) at Months 15, 18 and 24
Description: as for outcome 31
Time Frame: Baseline (Month 0) to Months 15, 18 and 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
ratio
  Baseline (Month 15): number analyzed (Participants) | 59 | 167
  Baseline (Month 15) | 1.409 (0.6706) | 1.440 (0.6714)
  Change from Baseline to Month 15: number analyzed (Participants) | 59 | 167
  Change from Baseline to Month 15 | 0.075 (0.5982) | 0.213 (0.6462)
  Baseline (Month 18): number analyzed (Participants) | 53 | 167
  Baseline (Month 18) | 1.389 (0.6699) | 1.440 (0.6895)
  Change from Baseline to Month 18: number analyzed (Participants) | 53 | 167
  Change from Baseline to Month 18 | 0.094 (0.5891) | 0.219 (0.5559)
  Baseline (Month 24): number analyzed (Participants) | 56 | 158
  Baseline (Month 24) | 1.426 (0.6841) | 1.444 (0.6838)
  Change from Baseline to Month 24: number analyzed (Participants) | 56 | 158
  Change from Baseline to Month 24 | 0.064 (0.8103) | 0.166 (0.6086)

33. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Hyaluronic Acid at Months 6 and 12
Description: Hyaluronic acid is a non-invasive hepatic fibrosis marker. A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline (Month 0) to Months 6 and 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
ng/mL
  Baseline (Month 6): number analyzed (Participants) | 128 | 128
  Baseline (Month 6) | 68.7 (107.63) | 68.2 (78.88)
  Change from Baseline to Month 6: number analyzed (Participants) | 128 | 128
  Change from Baseline to Month 6 | -2.4 (75.03) | 10.7 (79.58)
  Baseline (Month 12): number analyzed (Participants) | 122 | 121
  Baseline (Month 12) | 70.7 (110.49) | 69.5 (80.56)
  Change from Baseline to Month 12: number analyzed (Participants) | 122 | 121
  Change from Baseline to Month 12 | -0.2 (81.30) | 10.9 (58.46)

34. Secondary Outcome: Change From Baseline in Non-invasive Marker of Hepatic Fibrosis: Hyaluronic Acid at Months 18 and 24
Description: Hyaluronic acid is a non-invasive hepatic fibrosis marker. A positive change from Baseline indicates increased fibrosis.
Time Frame: Baseline (Month 0) to Months 18 and 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
ng/mL
  Baseline (Month 18): number analyzed (Participants) | 58 | 170
  Baseline (Month 18) | 46.4 (32.67) | 79.6 (111.36)
  Change from Baseline to Month 18: number analyzed (Participants) | 58 | 170
  Change from Baseline to Month 18 | 5.7 (34.66) | 1.4 (81.20)
  Baseline (Month 24): number analyzed (Participants) | 57 | 164
  Baseline (Month 24) | 46.6 (32.91) | 79.7 (112.46)
  Change from Baseline to Month 24: number analyzed (Participants) | 57 | 164
  Change from Baseline to Month 24 | 19.3 (70.64) | 13.0 (95.00)

35. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: Nonalcoholic Fatty Liver Disease (NAFLD) Fibrosis Score (NFS) at Months 3, 6 and 12
Description: NFS is calculated using formula: NFS = -1.675 + 0.037 * age (years) + 0.094 * Body mass index (BMI) (kg/m^2) + 1.13 * Impaired fasting glucose (IFG)/diabetes (yes = 1, no = 0) + 0.99 * Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) ratio - 0.013 × platelet (*10^9/L) - 0.66 * albumin (g/dL). A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline (Month 0) to Months 3, 6 and 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
ng/mL
  Baseline (Month 3): number analyzed (Participants) | 125 | 125
  Baseline (Month 3) | -1.227 (1.5255) | -1.012 (1.2558)
  Change from Baseline to Month 3: number analyzed (Participants) | 125 | 125
  Change from Baseline to Month 3 | 0.029 (0.5150) | 0.087 (0.4608)
  Baseline (Month 6): number analyzed (Participants) | 125 | 119
  Baseline (Month 6) | -1.119 (1.4935) | -1.064 (1.2403)
  Change from Baseline to Month 6: number analyzed (Participants) | 125 | 119
  Change from Baseline to Month 6 | 0.051 (0.4747) | 0.094 (0.5460)
  Baseline (Month 12): number analyzed (Participants) | 115 | 108
  Baseline (Month 12) | -1.132 (1.4609) | -1.040 (1.1393)
  Change from Baseline to Month 12: number analyzed (Participants) | 115 | 108
  Change from Baseline to Month 12 | 0.121 (0.5117) | 0.139 (0.5016)

36. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: NAFLD Fibrosis Score (NFS) at Months 15, 18 and 24
Description: as for outcome 35
Time Frame: Baseline (Month 0) to Months 15, 18 and 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
ng/mL
  Baseline (Month 15): number analyzed (Participants) | 59 | 158
  Baseline (Month 15) | -1.252 (1.4602) | -1.051 (1.3410)
  Change from Baseline to Month 15: number analyzed (Participants) | 59 | 158
  Change from Baseline to Month 15 | 0.057 (0.5981) | 0.225 (0.5654)
  Baseline (Month 18): number analyzed (Participants) | 53 | 158
  Baseline (Month 18) | -1.284 (1.4910) | -1.057 (1.3309)
  Change from Baseline to Month 18: number analyzed (Participants) | 53 | 158
  Change from Baseline to Month 18 | 0.046 (0.5809) | 0.196 (0.5583)
  Baseline (Month 24): number analyzed (Participants) | 54 | 147
  Baseline (Month 24) | -1.245 (1.4778) | -1.100 (1.3228)
  Change from Baseline to Month 24: number analyzed (Participants) | 54 | 147
  Change from Baseline to Month 24 | 0.046 (0.6188) | 0.185 (0.6184)

37. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: Enhanced Liver Fibrosis Test (ELF) Score at Months 6 and 12
Description: The markers of fibrosis assessed in this test comprised hyaluronic acid (CHA), tissue inhibitor of metalloproteinase (CTIMP1) and procollagen III N-terminal peptide (CP3NP); these are components of the extracellular matrix and basement sinusoidal membrane of the liver and are elevated during activation of the stellate cell. The ELF tests were performed on Centaur device and the composite score was calculated as follows: ELF score = 2.278 + 0.851 ln(CHA) + 0.751 ln (CP3NP) + 0.394 ln(CTIMP1). ELF score < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis. A negative change from Baseline indicates decreased fibrosis.
Time Frame: Baseline (Month 0) to Months 6 and 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
ng/mL
  Baseline (Month 6): number analyzed (Participants) | 125 | 125
  Baseline (Month 6) | -0.786 (0.7179) | -0.837 (0.7238)
  Change from Baseline to Month 6: number analyzed (Participants) | 125 | 125
  Change from Baseline to Month 6 | -0.022 (0.4901) | 0.060 (0.5228)
  Baseline (Month 12): number analyzed (Participants) | 116 | 118
  Baseline (Month 12) | -0.795 (0.7435) | -0.801 (0.7162)
  Change from Baseline to Month 12: number analyzed (Participants) | 116 | 118
  Change from Baseline to Month 12 | -0.064 (0.5602) | 0.041 (0.5727)

38. Secondary Outcome: Change From Baseline in Non-invasive Markers of Hepatic Fibrosis: Enhanced Liver Fibrosis Test (ELF) Score at Months 18 and 24
Description: as for outcome 37
Time Frame: Baseline (Month 0) to Months 18 and 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
ng/mL
  Baseline (Month 18): number analyzed (Participants) | 57 | 164
  Baseline (Month 18) | -0.931 (0.6387) | -0.758 (0.7307)
  Change from Baseline to Month 18: number analyzed (Participants) | 57 | 164
  Change from Baseline to Month 18 | -0.129 (0.6606) | -0.087 (0.6113)
  Baseline (Month 24): number analyzed (Participants) | 56 | 157
  Baseline (Month 24) | -0.940 (0.6587) | -0.765 (0.7127)
  Change from Baseline to Month 24: number analyzed (Participants) | 56 | 157
  Change from Baseline to Month 24 | -0.024 (0.7375) | 0.096 (0.6437)

39. Secondary Outcome: Change From Baseline in Biomarkers of Hepatocyte Apoptosis: Caspase Cleaved (CK-18 [M-30]) Levels and Total M-65 (CK-18 [M-65]) Levels at Months 3, 6 and 12
Description: Caspase-cleaved cytokeratin levels (CK18M30) and total M-65 (CK-18 [M-65]) were measured as biomarkers of hepatocyte apoptosis. A negative change from Baseline indicates decreased hepatocyte apoptosis.
Time Frame: Baseline (Month 0) to Months 3, 6 and 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 143 | 144
U/L
  Baseline (Month 3): number analyzed (Participants) | 115 | 119
  Baseline (Month 3) | 601.6 (431.77) | 594.2 (554.20)
  Change from Baseline to Month 3: number analyzed (Participants) | 115 | 119
  Change from Baseline to Month 3 | -56.4 (451.14) | -59.0 (485.76)
  Baseline (Month 6): number analyzed (Participants) | 105 | 107
  Baseline (Month 6) | 550.3 (360.64) | 552.9 (393.92)
  Change from Baseline to Month 6: number analyzed (Participants) | 105 | 107
  Change from Baseline to Month 6 | 10.6 (461.98) | -26.1 (512.88)
  Baseline (Month 12): number analyzed (Participants) | 107 | 101
  Baseline (Month 12) | 555.3 (356.28) | 567.9 (500.53)
  Change from Baseline to Month 12: number analyzed (Participants) | 107 | 101
  Change from Baseline to Month 12 | 99.7 (824.50) | 107.8 (830.28)

40. Secondary Outcome: Change From Baseline in Biomarkers of Hepatocyte Apoptosis: Caspase Cleaved (CK-18 [M-30]) Levels and Total M-65 (CK-18 [M-65]) Levels at Months 15, 18 and 24
Description: as for outcome 39
Time Frame: Baseline (Month 0) to Months 15, 18 and 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 72 | 215
U/L
  CK-18(M30), Baseline (Month 15): number analyzed (Participants) | 51 | 145
  CK-18(M30), Baseline (Month 15) | 570.8 (297.42) | 536.4 (459.06)
  CK-18(M30), Change from Baseline to Month 15: number analyzed (Participants) | 51 | 145
  CK-18(M30), Change from Baseline to Month 15 | -39.6 (287.44) | -13.3 (450.16)
  CK-18(M30), Baseline (Month 18): number analyzed (Participants) | 51 | 149
  CK-18(M30), Baseline (Month 18) | 578.8 (293.93) | 540.9 (453.90)
  CK-18(M30), Change from Baseline to Month 18: number analyzed (Participants) | 51 | 149
  CK-18(M30), Change from Baseline to Month 18 | 23.8 (402.98) | 57.3 (476.92)
  CK-18(M30), Baseline (Month 24): number analyzed (Participants) | 50 | 143
  CK-18(M30), Baseline (Month 24) | 575.4 (293.64) | 541.8 (462.29)
  CK-18(M30), Change from Baseline to Month 24: number analyzed (Participants) | 50 | 143
  CK-18(M30), Change from Baseline to Month 24 | -30.0 (369.60) | 39.7 (437.60)
  CK-18(M65), Baseline (Month 15): number analyzed (Participants) | 51 | 145
  CK-18(M65), Baseline (Month 15) | 772.7 (337.24) | 687.4 (404.83)
  CK-18(M65), Change from Baseline to Month 15: number analyzed (Participants) | 51 | 145
  CK-18(M65), Change from Baseline to Month 15 | 134.7 (534.46) | 88.6 (559.11)
  CK-18(M65), Baseline (Month 18): number analyzed (Participants) | 51 | 149
  CK-18(M65), Baseline (Month 18) | 777.8 (344.07) | 694.8 (401.88)
  CK-18(M65), Change from Baseline to Month 18: number analyzed (Participants) | 51 | 149
  CK-18(M65), Change from Baseline to Month 18 | 158.0 (732.63) | 181.5 (620.57)
  CK-18(M65), Baseline (Month 24): number analyzed (Participants) | 50 | 143
  CK-18(M65), Baseline (Month 24) | 770.2 (335.05) | 693.9 (409.88)
  CK-18(M65), Change from Baseline to Month 24: number analyzed (Participants) | 50 | 143
  CK-18(M65), Change from Baseline to Month 24 | 7.4 (570.92) | 124.9 (522.08)

41. Secondary Outcome: Change From Baseline in Weight at Months 3, 6 and 12
Description: A negative change from Baseline represents decreased weight.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: Safety Analysis Set Year 1 included all participants who received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analysis at both Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
kg
  Baseline (Month 3): number analyzed (Participants) | 133 | 138
  Baseline (Month 3) | 97.21 (22.368) | 95.59 (20.590)
  Change from Baseline to Month 3: number analyzed (Participants) | 133 | 138
  Change from Baseline to Month 3 | -0.50 (2.652) | -0.63 (2.632)
  Baseline (Month 6): number analyzed (Participants) | 130 | 132
  Baseline (Month 6) | 97.18 (22.224) | 95.18 (20.386)
  Change from Baseline to Month 6: number analyzed (Participants) | 130 | 132
  Change from Baseline to Month 6 | -0.55 (3.319) | -0.47 (3.466)
  Baseline (Month 12): number analyzed (Participants) | 126 | 122
  Baseline (Month 12) | 96.63 (22.139) | 95.06 (20.651)
  Change from Baseline to Month 12: number analyzed (Participants) | 126 | 122
  Change from Baseline to Month 12 | -0.08 (4.301) | -0.28 (4.166)

42. Secondary Outcome: Change From Baseline in Weight at Months 15, 18 and 24
Description: A negative change from Baseline represents decreased weight.
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: Safety Analysis Set Year 2 included all participants who received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analysis at both Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
kg
  Baseline (Month 15): number analyzed (Participants) | 59 | 174
  Baseline (Month 15) | 98.25 (24.087) | 95.32 (20.749)
  Change from Baseline to Month 15: number analyzed (Participants) | 59 | 174
  Change from Baseline to Month 15 | 0.15 (3.448) | -0.44 (4.257)
  Baseline (Month 18): number analyzed (Participants) | 58 | 173
  Baseline (Month 18) | 96.98 (22.210) | 95.23 (20.823)
  Change from Baseline to Month 18: number analyzed (Participants) | 58 | 173
  Change from Baseline to Month 18 | 0.05 (4.194) | -0.16 (4.458)
  Baseline (Month 24): number analyzed (Participants) | 58 | 166
  Baseline (Month 24) | 96.98 (22.210) | 95.19 (20.972)
  Change from Baseline to Month 24: number analyzed (Participants) | 58 | 166
  Change from Baseline to Month 24 | -0.91 (5.649) | -0.56 (5.081)

43. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Months 3, 6 and 12
Description: The body mass index is a value derived from the mass (weight in kgs) and height (in centimeters) of an individual and is calculated as the body mass divided by the square of the body height. A negative change from Baseline represents decreased BMI.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
kg/m^2
  Baseline (Month 3): number analyzed (Participants) | 133 | 135
  Baseline (Month 3) | 34.129 (7.2492) | 33.706 (5.7812)
  Change from Baseline to Month 3: number analyzed (Participants) | 133 | 135
  Change from Baseline to Month 3 | -0.172 (0.9200) | -0.232 (0.9500)
  Baseline (Month 6): number analyzed (Participants) | 130 | 129
  Baseline (Month 6) | 34.196 (7.3086) | 33.547 (5.6037)
  Change from Baseline to Month 6: number analyzed (Participants) | 130 | 129
  Change from Baseline to Month 6 | -0.182 (1.1558) | -0.196 (1.2500)
  Baseline (Month 12): number analyzed (Participants) | 126 | 119
  Baseline (Month 12) | 34.029 (7.1358) | 33.374 (5.6631)
  Change from Baseline to Month 12: number analyzed (Participants) | 126 | 119
  Change from Baseline to Month 12 | -0.013 (1.7507) | -0.145 (1.4891)

44. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Months 15, 18 and 24
Description: as for outcome 43
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
kg/m^2
  Baseline (Month 15): number analyzed (Participants) | 59 | 171
  Baseline (Month 15) | 34.713 (8.0431) | 33.392 (5.9669)
  Change from Baseline to Month 15: number analyzed (Participants) | 59 | 171
  Change from Baseline to Month 15 | -0.006 (1.2799) | -0.113 (1.6311)
  Baseline (Month 18): number analyzed (Participants) | 58 | 170
  Baseline (Month 18) | 34.473 (7.8964) | 33.345 (5.9443)
  Change from Baseline to Month 18: number analyzed (Participants) | 58 | 170
  Change from Baseline to Month 18 | -0.039 (1.5931) | -0.040 (1.7153)
  Baseline (Month 24): number analyzed (Participants) | 58 | 163
  Baseline (Month 24) | 34.473 (7.8964) | 33.278 (6.0012)
  Change from Baseline to Month 24: number analyzed (Participants) | 58 | 163
  Change from Baseline to Month 24 | -0.393 (2.0613) | -0.178 (1.8515)

45. Secondary Outcome: Change From Baseline in Waist Circumference at Months 3, 6 and 12
Description: A negative change from Baseline represents decreased in waist circumference.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
cm
  Baseline (Month 3): number analyzed (Participants) | 131 | 135
  Baseline (Month 3) | 110.35 (14.866) | 110.25 (13.406)
  Change from Baseline to Month 3: number analyzed (Participants) | 131 | 135
  Change from Baseline to Month 3 | 0.07 (5.147) | 0.05 (5.396)
  Baseline (Month 6): number analyzed (Participants) | 129 | 129
  Baseline (Month 6) | 110.42 (14.986) | 110.12 (13.561)
  Change from Baseline to Month 6: number analyzed (Participants) | 129 | 129
  Change from Baseline to Month 6 | 0.42 (8.827) | -0.54 (5.876)
  Baseline (Month 12): number analyzed (Participants) | 123 | 118
  Baseline (Month 12) | 109.77 (14.617) | 110.02 (13.711)
  Change from Baseline to Month 12: number analyzed (Participants) | 123 | 118
  Change from Baseline to Month 12 | 0.44 (6.584) | -1.10 (6.255)

46. Secondary Outcome: Change From Baseline in Waist Circumference at Months 15, 18 and 24
Description: A negative change from Baseline represents decreased in waist circumference.
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
cm
  Baseline (Month 15): number analyzed (Participants) | 57 | 172
  Baseline (Month 15) | 110.19 (14.360) | 110.26 (14.486)
  Change from Baseline to Month 15: number analyzed (Participants) | 57 | 172
  Change from Baseline to Month 15 | 0.52 (5.520) | -0.18 (6.280)
  Baseline (Month 18): number analyzed (Participants) | 56 | 170
  Baseline (Month 18) | 109.48 (12.703) | 110.25 (14.517)
  Change from Baseline to Month 18: number analyzed (Participants) | 56 | 170
  Change from Baseline to Month 18 | 1.36 (7.966) | -0.21 (6.578)
  Baseline (Month 24): number analyzed (Participants) | 58 | 163
  Baseline (Month 24) | 109.36 (12.608) | 110.08 (14.606)
  Change from Baseline to Month 24: number analyzed (Participants) | 58 | 163
  Change from Baseline to Month 24 | 0.11 (7.907) | -1.00 (6.503)

47. Secondary Outcome: Change From Baseline in Hip Circumference at Months 3, 6 and 12
Description: A negative change from Baseline represents decreased hip circumference.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
cm
  Baseline (Month 3): number analyzed (Participants) | 129 | 130
  Baseline (Month 3) | 114.92 (16.150) | 112.35 (13.802)
  Change from Baseline to Month 3: number analyzed (Participants) | 129 | 130
  Change from Baseline to Month 3 | -0.30 (4.921) | -0.11 (6.475)
  Baseline (Month 6): number analyzed (Participants) | 127 | 124
  Baseline (Month 6) | 115.09 (16.270) | 112.16 (13.320)
  Change from Baseline to Month 6: number analyzed (Participants) | 127 | 124
  Change from Baseline to Month 6 | -0.84 (4.396) | -0.18 (5.715)
  Baseline (Month 12): number analyzed (Participants) | 121 | 113
  Baseline (Month 12) | 114.46 (15.970) | 111.66 (13.376)
  Change from Baseline to Month 12: number analyzed (Participants) | 121 | 113
  Change from Baseline to Month 12 | -0.25 (5.876) | -0.08 (7.474)

48. Secondary Outcome: Change From Baseline in Hip Circumference at Months 15, 18 and 24
Description: A negative change from Baseline represents decreased hip circumference.
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
cm
  Baseline (Month 15): number analyzed (Participants) | 58 | 165
  Baseline (Month 15) | 114.56 (17.500) | 113.00 (14.183)
  Change from Baseline to Month 15: number analyzed (Participants) | 58 | 165
  Change from Baseline to Month 15 | -0.06 (5.361) | -0.83 (7.050)
  Baseline (Month 18): number analyzed (Participants) | 55 | 162
  Baseline (Month 18) | 114.28 (17.871) | 112.70 (14.168)
  Change from Baseline to Month 18: number analyzed (Participants) | 55 | 162
  Change from Baseline to Month 18 | 0.55 (7.791) | -0.90 (6.066)
  Baseline (Month 24): number analyzed (Participants) | 58 | 157
  Baseline (Month 24) | 114.34 (17.408) | 112.88 (14.225)
  Change from Baseline to Month 24: number analyzed (Participants) | 58 | 157
  Change from Baseline to Month 24 | -0.95 (7.700) | -1.21 (6.677)

49. Secondary Outcome: Change From Baseline in Forearm Circumference at Months 3, 6 and 12
Description: A negative change from Baseline represents decreased forearm circumference.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
cm
  Baseline (Month 3): number analyzed (Participants) | 127 | 132
  Baseline (Month 3) | 32.95 (7.346) | 33.38 (4.835)
  Change from Baseline to Month 3: number analyzed (Participants) | 127 | 132
  Change from Baseline to Month 3 | 0.97 (6.023) | 0.10 (6.486)
  Baseline (Month 6): number analyzed (Participants) | 126 | 126
  Baseline (Month 6) | 32.70 (7.290) | 33.25 (4.734)
  Change from Baseline to Month 6: number analyzed (Participants) | 126 | 126
  Change from Baseline to Month 6 | 0.82 (6.748) | -0.01 (3.447)
  Baseline (Month 12): number analyzed (Participants) | 120 | 115
  Baseline (Month 12) | 32.51 (7.277) | 33.09 (4.771)
  Change from Baseline to Month 12: number analyzed (Participants) | 120 | 115
  Change from Baseline to Month 12 | 0.83 (6.656) | -0.43 (3.516)

50. Secondary Outcome: Change From Baseline in Forearm Circumference at Months 15, 18 and 24
Description: A negative change from Baseline represents decreased forearm circumference.
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
cm
  Baseline (Month 15): number analyzed (Participants) | 57 | 168
  Baseline (Month 15) | 32.88 (7.783) | 32.91 (5.662)
  Change from Baseline to Month 15: number analyzed (Participants) | 57 | 168
  Change from Baseline to Month 15 | 1.61 (6.534) | 0.01 (5.052)
  Baseline (Month 18): number analyzed (Participants) | 55 | 166
  Baseline (Month 18) | 32.63 (7.718) | 32.87 (5.696)
  Change from Baseline to Month 18: number analyzed (Participants) | 55 | 166
  Change from Baseline to Month 18 | 1.79 (6.715) | 0.02 (4.709)
  Baseline (Month 24): number analyzed (Participants) | 57 | 159
  Baseline (Month 24) | 32.79 (7.660) | 33.02 (5.561)
  Change from Baseline to Month 24: number analyzed (Participants) | 57 | 159
  Change from Baseline to Month 24 | 0.78 (6.124) | -0.64 (4.408)

51. Secondary Outcome: Change From Baseline in Tricep Skinfold Thickness at Months 3, 6 and 12
Description: A negative change from Baseline represents decreased Tricep Skinfold Thickness.
Time Frame: Baseline (Day 1) to Months 3, 6 and 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 144 | 144
mm
  Baseline (Month 3): number analyzed (Participants) | 127 | 131
  Baseline (Month 3) | 28.32 (13.677) | 25.41 (12.593)
  Change from Baseline to Month 3: number analyzed (Participants) | 127 | 131
  Change from Baseline to Month 3 | -1.21 (6.548) | -0.62 (8.704)
  Baseline (Month 6): number analyzed (Participants) | 128 | 125
  Baseline (Month 6) | 28.53 (13.763) | 25.38 (12.769)
  Change from Baseline to Month 6: number analyzed (Participants) | 128 | 125
  Change from Baseline to Month 6 | -2.72 (8.091) | -1.52 (9.287)
  Baseline (Month 12): number analyzed (Participants) | 122 | 115
  Baseline (Month 12) | 28.54 (13.981) | 25.14 (12.969)
  Change from Baseline to Month 12: number analyzed (Participants) | 122 | 115
  Change from Baseline to Month 12 | -1.34 (9.389) | -0.26 (10.653)

52. Secondary Outcome: Change From Baseline in Tricep Skinfold Thickness at Months 15, 18 and 24
Description: A negative change from Baseline represents decreased Tricep Skinfold Thickness.
Time Frame: Baseline (Day 1) to Months 15, 18 and 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | CVC 150 mg
Number analyzed (Participants) | 60 | 182
mm
  Baseline (Month 15): number analyzed (Participants) | 57 | 170
  Baseline (Month 15) | 29.84 (14.422) | 25.41 (13.212)
  Change from Baseline to Month 15: number analyzed (Participants) | 57 | 170
  Change from Baseline to Month 15 | -1.45 (9.364) | -1.59 (8.918)
  Baseline (Month 18): number analyzed (Participants) | 55 | 168
  Baseline (Month 18) | 29.84 (14.655) | 25.07 (12.856)
  Change from Baseline to Month 18: number analyzed (Participants) | 55 | 168
  Change from Baseline to Month 18 | -2.27 (8.854) | -2.64 (8.864)
  Baseline (Month 24): number analyzed (Participants) | 56 | 160
  Baseline (Month 24) | 29.91 (14.532) | 24.82 (13.025)
  Change from Baseline to Month 24: number analyzed (Participants) | 56 | 160
  Change from Baseline to Month 24 | -3.11 (8.553) | -1.33 (10.521)

ADVERSE EVENTS:
Time Frame: Baseline to Year 2
Description: Safety Analysis Set Year 1 and Year 2 included all participants who received at least 1 dose of study drug.
Arm/Group | CVC 150mg/CVC 150 mg | Placebo/Cenicriviroc (CVC) 150 mg | Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 25/144 | 8/72 | 12/72
Other Adverse Events (participants affected / at risk) | 127/144 | 59/72 | 60/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVC 150mg/CVC 150 mg (N=144) | Placebo/Cenicriviroc (CVC) 150 mg (N=72) | Placebo/Placebo (N=72)
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Peripheral nerve sheath tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vasculitis gastrointestinal (Gastrointestinal disorders) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Bladder dysplasia (Renal and urinary disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVC 150mg/CVC 150 mg (N=144) | Placebo/Cenicriviroc (CVC) 150 mg (N=72) | Placebo/Placebo (N=72)
Diarrhoea (Gastrointestinal disorders) | 32 | 14 | 15
Abdominal pain upper (Gastrointestinal disorders) | 16 | 12 | 10
Abdominal pain (Gastrointestinal disorders) | 18 | 6 | 11
Nausea (Gastrointestinal disorders) | 28 | 6 | 8
Abdominal distension (Gastrointestinal disorders) | 13 | 4 | 0
Constipation (Gastrointestinal disorders) | 13 | 4 | 6
Flatulence (Gastrointestinal disorders) | 9 | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 3 | 4
Vomiting (Gastrointestinal disorders) | 18 | 3 | 5
Fatigue (General disorders) | 24 | 10 | 13
Oedema peripheral (General disorders) | 5 | 5 | 3
Pyrexia (General disorders) | 8 | 4 | 1
Urinary tract infection (Infections and infestations) | 17 | 10 | 4
Nasopharyngitis (Infections and infestations) | 21 | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 18 | 9 | 8
Influenza (Infections and infestations) | 11 | 3 | 3
Sinusitis (Infections and infestations) | 18 | 3 | 9
Ear infection (Infections and infestations) | 5 | 2 | 4
Bronchitis (Infections and infestations) | 10 | 1 | 7
Gastroenteritis (Infections and infestations) | 3 | 1 | 4
Procedural pain (Injury, poisoning and procedural complications) | 5 | 2 | 9
Alanine aminotransferase increased (Investigations) | 15 | 9 | 5
Blood creatine phosphokinase increased (Investigations) | 3 | 5 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 | 5 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 1 | 6
Headache (Nervous system disorders) | 24 | 15 | 9
Dizziness (Nervous system disorders) | 13 | 0 | 5
Insomnia (Psychiatric disorders) | 10 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 12 | 3 | 8
Hypertension (Vascular disorders) | 10 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.